CLINICAL TRIAL: NCT04263896
Title: Bowel Function After Minimally Invasive Hysterectomy: A Randomized Controlled Trial
Brief Title: Bowel Function After Minimally Invasive Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB19-0436
Record Dates: First submitted 2019-08-29; First posted 2020-02-11 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-06

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350

STUDY DESIGN:
Intervention Model Description: Following enrollment subjects will be randomized into the intervention/treatment arm and control arm through a randomizing process in the investigator's database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Participants receiving pre-operative laxative (Experimental): Participants will receive 10 doses, 17g each, of polyethylene glycol 3350. They will be instructed to take 1 dose/packet each day for 10 days leading up to their surgery.
  Interventions: Drug: Polyethylene Glycol 3350
- Participants not receiving pre-operative laxative (No Intervention): Participants will not be given any laxatives.

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — Participants will take 1 17g pack per day for 10 days preceding surgery.
  Other Names: Miralax
  Arms: Participants receiving pre-operative laxative

SUMMARY:
Postoperative constipation affects up to a third of women undergoing minimally invasive (MIS) gynecologic surgery and is a major source of anxiety and discomfort. The average time to first bowel movement after gynecologic surgery is about 2 to 4 days and some factors responsible for this include anesthesia inhibitory effect on gastrointestinal motility, opioid pain medication use, chronic nonsteroidal anti-inflammatory drugs (NSAID) use and anatomic manipulation.

There are no established regimens to manage postoperative constipation after minimally invasive gynecologic surgery. Two studies evaluating the implementation of postoperative bowel regimen with polyethylene glycol (PEG) and with Senna and Docusate found no significant impact on postoperative bowel function. There have been no studies looking at the effect of preoperative bowel regimens on postoperative bowel function.

The purpose of this study is to evaluate postoperative bowel function after minimally invasive hysterectomy in women receiving a preoperative 10-day bowel regimen of PEG daily.

DETAILED DESCRIPTION:
Following enrollment subjects will be randomized into the intervention/treatment arm and control arm. All subjects will be asked to complete a baseline demographic form and three questionnaires (Patient Assessment of Constipation Symptoms (PAC-SYM), Patient Assessment of Constipation Quality of Life (PAC- QOL), Wexner Constipation score). Additional demographic information will be obtained from chart review. This information will include past medical history, use of constipating medications, use of daily pain medications, chronic pain history, use of daily fiber supplementation.

Subjects in the intervention arm will be given 10-day supply of Miralax and instructed on its use. They will take this medication for the 10 days prior to surgery. Subjects in the control arm will continue with standard care prior to surgery.

Post operatively, all subjects will complete a diary for 7 days. In this diary they will record details about their bowel movements (time of movement, discomfort, texture of stool). They will also report average daily pain levels ( with a visual analog scale), daily pain medication use (time, medication, total number of pills).

At the end of the 7th day all subjects will complete the same PAC questionnaires as they did pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Any woman ≥ 18 years of age undergoing a minimally invasive hysterectomy (Laparoscopic, robotic, vaginal)
* Able to understand the consenting process and willing to participate in study

Exclusion Criteria:

* Planned laparotomy
* Emergent surgery
* Regular preoperative use of PEG 3350, laxatives, enemas or suppositories
* Planned bowel surgery
* Presence of colostomy
* Inability to consent
* Medical problems as follows:
* Chronic Kidney Disease (Cr: > 1.2 mg/dL)
* Insulin-Dependent Diabetes Mellitus
* Cardiac disease
* Gastric ulcers
* Difficulty swallowing or esophageal stricture
* Persistent nausea or vomiting
* Signs or symptoms of a small bowel obstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Glass, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel M, Schimpf MO, O'Sullivan DM, LaSala CA. The use of senna with docusate for postoperative constipation after pelvic reconstructive surgery: a randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol. 2010 May;202(5):479.e1-5. doi: 10.1016/j.ajog.2010.01.003. Epub 2010 Mar 6. PMID 20207340
- [Result] Edenfield AL, Siddiqui NY, Wu JM, Dieter AA, Garrett MA, Visco AG. Polyethylene Glycol 3350 and Docusate Sodium Compared With Docusate Sodium Alone After Urogynecologic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2016 Sep;128(3):543-9. doi: 10.1097/AOG.0000000000001565. PMID 27500338
- [Result] Clarke A, Black N, Rowe P, Mott S, Howle K. Indications for and outcome of total abdominal hysterectomy for benign disease: a prospective cohort study. Br J Obstet Gynaecol. 1995 Aug;102(8):611-20. doi: 10.1111/j.1471-0528.1995.tb11398.x. PMID 7654638
- [Result] Mythen MG. Postoperative gastrointestinal tract dysfunction: an overview of causes and management strategies. Cleve Clin J Med. 2009 Nov;76 Suppl 4:S66-71. doi: 10.3949/ccjm.76.s4.11. PMID 19880839
- [Result] Pappagallo M. Incidence, prevalence, and management of opioid bowel dysfunction. Am J Surg. 2001 Nov;182(5A Suppl):11S-18S. doi: 10.1016/s0002-9610(01)00782-6. PMID 11755892
- [Result] Iwanoff C, Giannopoulos M, Salamon C. Follow-up postoperative calls to reduce common postoperative complaints among urogynecology patients. Int Urogynecol J. 2019 Oct;30(10):1667-1672. doi: 10.1007/s00192-018-3809-x. Epub 2018 Nov 9. PMID 30413866
- [Result] Caljouw MA, Hogendorf-Burgers ME. GYNOTEL: telephone advice to gynaecological surgical patients after discharge. J Clin Nurs. 2010 Dec;19(23-24):3301-6. doi: 10.1111/j.1365-2702.2010.03395.x. Epub 2010 Oct 14. PMID 20946445
- [Result] Spence-Jones C, Kamm MA, Henry MM, Hudson CN. Bowel dysfunction: a pathogenic factor in uterovaginal prolapse and urinary stress incontinence. Br J Obstet Gynaecol. 1994 Feb;101(2):147-52. doi: 10.1111/j.1471-0528.1994.tb13081.x. PMID 8305390
- [Result] Arya LA, Novi JM, Shaunik A, Morgan MA, Bradley CS. Pelvic organ prolapse, constipation, and dietary fiber intake in women: a case-control study. Am J Obstet Gynecol. 2005 May;192(5):1687-91. doi: 10.1016/j.ajog.2004.11.032. PMID 15902178
- [Result] Ramirez PT, Klemer DP. Vaginal evisceration after hysterectomy: a literature review. Obstet Gynecol Surv. 2002 Jul;57(7):462-7. doi: 10.1097/00006254-200207000-00023. PMID 12172223
- [Result] Hur HC, Lightfoot M, McMillin MG, Kho KA. Vaginal cuff dehiscence and evisceration: a review of the literature. Curr Opin Obstet Gynecol. 2016 Aug;28(4):297-303. doi: 10.1097/GCO.0000000000000294. PMID 27310715
- [Result] McNanley A, Perevich M, Glantz C, Duecy EE, Flynn MK, Buchsbaum G. Bowel function after minimally invasive urogynecologic surgery: a prospective randomized controlled trial. Female Pelvic Med Reconstr Surg. 2012 Mar-Apr;18(2):82-5. doi: 10.1097/SPV.0b013e3182455529. PMID 22453316
- [Result] Marciniak CM, Toledo S, Lee J, Jesselson M, Bateman J, Grover B, Tierny J. Lubiprostone vs Senna in postoperative orthopedic surgery patients with opioid-induced constipation: a double-blind, active-comparator trial. World J Gastroenterol. 2014 Nov 21;20(43):16323-33. doi: 10.3748/wjg.v20.i43.16323. PMID 25473191
- [Result] Iyigun E, Ayhan H, Demircapar A, Tastan S. Impact of preoperative defecation pattern on postoperative constipation for patients undergoing cardiac surgery. J Clin Nurs. 2017 Feb;26(3-4):495-501. doi: 10.1111/jocn.13473. Epub 2016 Aug 15. PMID 27404560
- [Result] Dipalma JA, Cleveland MV, McGowan J, Herrera JL. A randomized, multicenter, placebo-controlled trial of polyethylene glycol laxative for chronic treatment of chronic constipation. Am J Gastroenterol. 2007 Jul;102(7):1436-41. doi: 10.1111/j.1572-0241.2007.01199.x. Epub 2007 Mar 31. PMID 17403074
- [Result] Yiannakou Y, Tack J, Piessevaux H, Dubois D, Quigley EMM, Ke MY, Da Silva S, Joseph A, Kerstens R. The PAC-SYM questionnaire for chronic constipation: defining the minimal important difference. Aliment Pharmacol Ther. 2017 Dec;46(11-12):1103-1111. doi: 10.1111/apt.14349. Epub 2017 Oct 6. PMID 28983926
- [Result] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Not Receiving Pre-operative Laxative: Participants will not be given any laxatives prophylactically, and will follow all standard of care pre-surgical instructions
Period: Overall Study
Arm/Group | Participants Receiving Pre-operative Laxative | Participants Not Receiving Pre-operative Laxative
Started | 50 | 47
Completed | 33 | 28
Not Completed | 17 | 19
Not completed — Withdrawal by Subject | 2 | 4
Not completed — converted to open procedure | 0 | 1
Not completed — Lost to Follow-up | 9 | 11
Not completed — surveys lost in mail | 5 | 3
Not completed — excluded from analysis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Not Receiving Pre-operative Laxative: Participants will not be given any pre-operative laxatives either through the study or through standard of care.
- Total: Total of all reporting groups
Arm/Group | Participants Receiving Pre-operative Laxative | Participants Not Receiving Pre-operative Laxative | Total
Number analyzed (Participants) | 33 | 28 | 61
Age, Continuous [Mean (Standard Deviation); unit: year] | 44 (10.4) | 48.1 (10) | 46 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Patient Assessment of Constipation Symptoms Questionnaire (PAC-SYM) Score
Description: Constipation will be evaluated both preoperatively and postoperatively using a validated questionnaires (PAC-SYM/PAC-QOL). Patient assessment of constipation symptoms (PAC-SYM) - The Patient Assessment of Constipation-Symptoms (PAC-SYM) questionnaire, developed through psychometric evaluation of adults with chronic constipation, is a tool for assessing the severity of patient-reported symptoms of this disorder. The 12-item questionnaire is divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom burden.
Time Frame: change in score from 10 days pre-operation to 7 days post-operation
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Participants Receiving Pre-operative Laxative | Participants Not Receiving Pre-operative Laxative
Number analyzed (Participants) | 24 | 27
score | 1.1 (0.7) | 0.6 (0.6)

2. Primary Outcome: Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) Score
Description: Patient assessment of constipation quality of life (PAC-QOL) - PAC-Qol is a self-reported questionnaire, was used to measure the quality of life of patients.9 The validated PAC-QoL is composed of 28 items grouped into four subscales: physical discomfort, psychosocial discomfort, worries and concerns, and satisfaction. The first three subscales are used to assess the patient dissatisfaction index, with an overall score ranging from 0 to 96 (where lower scores correspond to better quality of life). The satisfaction subscale includes four items with a global score ranging from 0 to 16, so that each patient's self-reported definitive outcome is defined as either poor (0-4), fairly good (5-8), good (9-12), or excellent (13-16).
Time Frame: change in score from 10 days pre-operation to 7 days post-operation
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Participants Receiving Pre-operative Laxative | Participants Not Receiving Pre-operative Laxative
Number analyzed (Participants) | 23 | 27
score
  Satisfaction | 8.4 (4.7) | 10 (4.2)
  Dissatisfaction | 21.6 (19.7) | 16.5 (14.9)

3. Secondary Outcome: Visual Analog Scale for Pain Management
Description: Visual analog scale - The visual analog scale (VAS) is a measure of subjective pain intensity. It is a continuous scale comprised of a horizontal visual analog scale that is 100 mm in length. The subject will place a mark on the scale to indicate the intensity of her pain. 0 mm would be no pain, 100 mm would be the greatest imaginable pain. Any mark in between will be measured in mm to indicate degree of pain the subject is experiencing.
Time Frame: The 7 days after surgery (surgery is D0)
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Participants Receiving Pre-operative Laxative | Participants Not Receiving Pre-operative Laxative
Number analyzed (Participants) | 33 | 28
score
  Day 1 | 5.807692 (2.112235) | 5.934615 (2.158507)
  day 2 | 5.114815 (1.886736) | 5.516 (1.993517)
  Day 3 | 4.572 (1.943691) | 4.681481 (2.068451)
  Day 4 | 3.919231 (2.234461) | 3.91 (1.659694)
  Day 5 | 3.580769 (2.249092) | 3.902692 (2.076619)
  Day 6 | 3.494 (2.386434) | 3.193478 (1.949843)
  Day 7 | 3.1044 (2.345364) | 3.153846 (2.423919)

4. Secondary Outcome: Pain Medication Consumption Tracking by Participant
Description: Dosages of pain medication consumption will be collected for up to 7 days post-surgery.
Time Frame: The 7 days after surgery (surgery is D0)
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Participants Receiving Pre-operative Laxative | Participants Not Receiving Pre-operative Laxative
Number analyzed (Participants) | 33 | 28
morphine milligram equivalents
  day 1 | 11.82692 (8.903867) | 14.33333 (13.11312)
  day 2 | 8.981481 (9.982178) | 12.58333 (15.51533)
  Day 3 | 7.410714 (9.824434) | 7.758621 (12.0702)
  Day 4 | 4.017857 (9.362536) | 5 (10.48809)
  Day 5 | 2.222222 (5.814989) | 2.258065 (4.625781)
  Day 6 | 1.388889 (3.126602) | 0.8333333 (2.653343)
  Day 7 | 1.388889 (3.126602) | 0.483871 (1.981093)

5. Secondary Outcome: Wexner/ Constipation Scoring System/1996 Cleveland Clinic Score / Agachan Score
Description: Wexner a commonly used scoring system, is designed to assess the prevalence and severity of constipation. It is based on pathophysiological definition of constipation. The scoring system is based on eight variables (frequency of bowel movements; difficult or painful evacuation; completeness of evacuation; abdominal pain; time per attempt; type of assistance including laxatives; digitations or enemas; number of unsuccessful attempts at evacuation in a 24-h period and duration of constipation). The CSS consists of seven items that are scored using a five-point Likert scale that ranges from 0 (none of the time) to 4 (all of the time) and one item that is rated on a 0-2 scale. A total score can range from 0 (normal) to 30 (severe constipation). A cutoff score of 15 suggests constipation.
Time Frame: 7 days before surgery
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Participants Receiving Pre-operative Laxative | Participants Not Receiving Pre-operative Laxative
Number analyzed (Participants) | 32 | 29
score | 7.3 (5) | 5.6 (3.7)

ADVERSE EVENTS:
Time Frame: two weeks
Description: There were no adverse events reported in this study
Arm/Group | Participants Receiving Pre-operative Laxative | Participants Not Receiving Pre-operative Laxative
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/28
Other Adverse Events (participants affected / at risk) | 0/33 | 0/28

LIMITATIONS AND CAVEATS:
Limitations of this study include a greater than expected dropout rate. With an anticipated 20% drop-out rate, we planned to include 80 patients in our statistical analysis. However, only 50-65 patients (depending on the outcome measure) had completed enough of the study materials to be included in the analysis, so our conclusions are under-powered. Furthermore, this was a non-blinded study, which may have contributed to a reporting bias among participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT04263896/Prot_SAP_001.pdf